CLINICAL TRIAL: NCT02224118
Title: Safety, Pharmacokinetics, and Pharmacodynamics of a Single Subcutaneous Dose of CNTO 3649 in Healthy Adult Men and Multiple Subcutaneous Doses of CNTO 3649 in Patients With Type 2 Diabetes Mellitus
Brief Title: Safety, Pharmacokinetics, and Pharmacodynamics Study of Single Dose of CNTO 3649 in Healthy Adult Men and Multiple Doses of CNTO 3649 in Participants With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR016429; JNS030-JPN-01 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2014-08-21; First posted 2014-08-25 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Healthy; Diabetes Mellitus, Type 2
Keywords: Healthy; Diabetes Mellitus, Type 2; CNTO 3649
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- CNTO 3649 10 mcg/kg (single dose) (Experimental): A single dose of 10 microgram per kilogram (mcg/kg) of CNTO 3649 will be administered as subcutaneous injection to healthy adult Japanese men.
  Interventions: Drug: CNTO 3649 10 mcg/kg
- CNT0 3649 30 mcg/kg (single dose) (Experimental): A single dose of 30 mcg/kg of CNTO 3649 will be administered as subcutaneous injection to healthy adult Japanese men.
  Interventions: Drug: CNT0 3649 30 mcg/kg
- CNTO 3649 100 mcg/kg (single dose) (Experimental): A single dose of 100 mcg/kg of CNTO 3649 will be administered as subcutaneous injection to healthy adult Japanese men.
  Interventions: Drug: CNTO 3649 100 mcg/kg
- CNTO 3649 300 mcg/kg (single dose) (Experimental): A single dose of 300 microgram per kilogram (mcg/kg) of CNTO 3649 will be administered as subcutaneous injection to healthy adult Japanese men.
  Interventions: Drug: CNTO 3649 300 mcg/kg
- CNT0 3649 30 mcg/kg (multiple dose) (Experimental): Participants with type 2 diabetes mellitus will be administered 30 mcg/kg CNTO 3649 as subcutaneous injection once a week for 4 weeks.
  Interventions: Drug: CNT0 3649 30 mcg/kg
- CNTO 3649 100 mcg/kg (multiple dose) (Experimental): Participants with type 2 diabetes mellitus will be administered 100 mcg/kg CNTO 3649 as subcutaneous injection once a week for 4 weeks.
  Interventions: Drug: CNTO 3649 100 mcg/kg
- Placebo (Placebo Comparator): Matching placebo to CNTO 3649 will be administered to both healthy volunteers and participants with type 2 diabetes mellitus.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CNTO 3649 10 mcg/kg — A single dose of 10 mcg/kg of CNTO 3649 will be administered as subcutaneous injection to healthy adult Japanese men.
  Arms: CNTO 3649 10 mcg/kg (single dose)
Drug: CNT0 3649 30 mcg/kg — A single dose of 30 mcg/kg of CNTO 3649 will be administered as subcutaneous injection to healthy adult Japanese men and multiple doses of 30 mcg/kg of CNTO 3649 will be administered to participants with type 2 diabetes mellitus as subcutaneous injections once weekly for 4 weeks.
  Arms: CNT0 3649 30 mcg/kg (multiple dose); CNT0 3649 30 mcg/kg (single dose)
Drug: CNTO 3649 100 mcg/kg — A single dose of 100 mcg/kg of CNTO 3649 will be administered as subcutaneous injection to healthy adult Japanese men and multiple doses of 100 mcg/kg of CNTO 3649 will be administered to participants with type 2 diabetes mellitus as subcutaneous injections once weekly for 4 weeks.
  Arms: CNTO 3649 100 mcg/kg (multiple dose); CNTO 3649 100 mcg/kg (single dose)
Drug: CNTO 3649 300 mcg/kg — A single dose of 300 mcg/kg of CNTO 3649 will be administered as subcutaneous injection to healthy adult Japanese men.
  Arms: CNTO 3649 300 mcg/kg (single dose)
Drug: Placebo — Matching Placebo to CNTO 3649 will be administered to both healthy volunteers and participants with type 2 diabetes mellitus.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the safety (adverse events, weight, blood pressure, pulse rate, body temperature, abdominal ultrasonography, standard 12-lead electrocardiography, and laboratory tests) of CNTO 3649 when administered once by subcutaneous injection in healthy adult Japanese men or once a week for 4 weeks in Japanese participants with type 2 diabetes mellitus (disorder in which there is decreased insulin in the body or the body's insulin is not effective, resulting in high blood sugar, increased thirst and urine, and many other side effects).

DETAILED DESCRIPTION:
This is a Phase 1, multi-arm and open-label (all knew the intervention of study) study to explore the safety, pharmacodynamics (the study of how drugs act on the body) and pharmacokinetics (the study of the way a drug enters and leaves the blood and tissues over time) of CNTO 3649. The study has been divided in Part 1 and 2. Part 1 includes healthy adult Japanese men and Part 2 includes Japanese participants with type 2 diabetes mellitus. The healthy adult Japanese men in part 1 will receive a single dose of either 10, 30, 100 or 300 microgram/milliliter (mcg/mL) of CNTO 3649 and participants in part 2 will receive subcutaneous doses of either 30 or 100 mcg/mL of CNTO 3649 once a week for 4 weeks. The study will have a Screening period of 28 days for Part 1 and 42 days for Part 2. Participants will primarily be assessed for safety (adverse events, weight, blood pressure, pulse rate, body temperature, abdominal ultrasonography, standard 12-lead electrocardiography, and laboratory test). The total duration of study will be 57 days for Part 1 and 92 days for Part 2.

ELIGIBILITY:
Inclusion Criteria:

Part 1

* Weighs greater than or equal to (>=) 50 kilogram (kg) and less than (<) 100 kg and has a body mass index (BMI) of >= 18.5 and <25.0 at the time of screening tests
* Is a non-smoker, or is able to refrain from smoking from 2 days before screening tests until completion of post-treatment examinations or follow-up investigations
* Is able to refrain from consuming alcohol from 2 days before screening tests until completion of screening tests, from 2 days before hospitalization (Day -4) until after discharge (Day 8), from 2 days before clinic visits (Days 13 and 20) until completion of tests at clinic visits (Days 15 and 22), and from 2 days before post-treatment examinations or follow-up investigations until completion of post-treatment examinations or follow-up investigations
* Has agreed to use a medically acceptable form of contraception (example [eg], condoms) from the day of hospitalization (Day -2) until completion of post-treatment examinations or follow-up investigations
* Has no clinically problematic abnormalities in medical examinations and tests before study treatment

Part 2

* Weighs >= 50 kg and <100 kg and has a BMI of >=18.5 and <37.0 at the time of screening tests
* Was diagnosed with type 2 diabetes mellitus at least 3 months before screening tests and this is being stably managed with dietary modification, exercise therapy, or sulfonylureas or biguanides If sulfonylureas or biguanides are being used, these have been used at a fixed dosage to stably manage the disease since at least 3 months before screening tests
* If the participant has hyperlipidemia, this has been stably managed with antihyperlipidemic drugs at a fixed dosage since at least 3 months before screening tests
* If the participant has hypertension, this has been stably managed with antihypertensive drugs at a fixed dosage since at least 3 months before screening tests
* Is a non-smoker, or is able to refrain from smoking during the hospitalization period and from 1 day before clinic visit days until completion of tests

Exclusion Criteria:

Part 1

* Has or has had hepatic, renal, central nervous system (including psychiatric), cardiovascular, respiratory, gastrointestinal, hematopoietic, ophthalmic, infectious, or endocrine disease that would make the participant unsuitable as a study participant
* Has had a malignant tumor within 5 years before study treatment
* Has undergone surgery that would make the participant unsuitable as a study participant within 12 weeks before screening tests
* Has or had acute disease that occurred within 7 days before study treatment
* Has or has had an eating disorder (pathological anorexia or bulimia)

Part 2

* If only dietary modification and exercise therapy are being used, fasting blood glucose is <130 milligram per deciliters (mg/dL) or >= 270 mg/dL in screening tests and at hospitalization (Day -1). If oral antihyperglycemic drugs are being used, fasting blood glucose is <100 mg/dL or >= 240 mg/dL at the time of screening tests and <120 mg/dL or >= 270 mg/dL at hospitalization (Day -1)
* If only dietary modification and exercise therapy are being used, HbA 1C at the time of Screening tests is <6% or >= 10 percent (%). If oral antihyperglycemic drugs are being used, HbA 1C at the time of screening tests is <6% or >=9%
* Has blood pressure or a pulse rate that is outside of the following ranges, or has hypertension and blood pressure or a pulse rate that is outside of the following ranges despite taking an antihypertensive drug at the same dosage since at least 3 months before screening tests
* Has or has had type 1 diabetes mellitus
* Has or has had autoimmune diabetes mellitus

Ages: 20 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2009-07; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants Reporting Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs) | Day 1 to 57 for CNTO 3649 10, 30, 100 and 300 mcg/kg (Part 1) or Day 1 to 92 for CNTO 3649 30 and 100 mcg/kg (Part 2)
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between administration of study drug and up to 57 for CNTO 3649 10, 30, 100 and 300 microgram per kilogram (mcg/kg) (Part 1); Day 1 to 92 for CNTO 3649 30 and 100 mcg/kg (Part 2) that would be absent before treatment or that may worsen relative to pre-treatment state.

SECONDARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) | Day 1 to 57 for CNTO 3649 10, 30, 100 and 300 mcg/kg (Part 1) or Day 1 to 92 for CNTO 3649 30 and 100 mcg/kg (Part 2)
  Maximum Observed Serum Concentration (Cmax) will be observed.
Time to Reach Maximum Observed Serum Concentration (Tmax) | Day 1 to 57 for CNTO 3649 10, 30, 100 and 300 mcg/kg (Part 1) or Day 1 to 92 for CNTO 3649 30 and 100 mcg/kg (Part 2)
  Time to Reach Maximum Observed Serum Concentration (Tmax) will be observed.
Terminal Phase Elimination Half Life (t1/2) | Day 1 to 57 for CNTO 3649 10, 30, 100 and 300 mcg/kg (Part 1) or Day 1 to 92 for CNTO 3649 30 and 100 mcg/kg (Part 2)
  Terminal phase elimination half-life is the time measured for the serum concentration to decrease by one half.
Area Under the Serum Concentration Time Curve From Time Zero to Last Measurable Concentration (AUC[0 - last]) | Day 1 to 57 for CNTO 3649 10, 30, 100 and 300 mcg/kg (Part 1) or Day 1 to 92 for CNTO 3649 30 and 100 mcg/kg (Part 2)
  Area Under the Serum Concentration Time Curve From Time Zero to Last Measurable Concentration (AUC[0 - last]) will be observed.
Area Under the Concentration-time Curve From Zero to Infinity (AUC [0 - infinity]) | Day 1 to 57 for CNTO 3649 10, 30, 100 and 300 mcg/kg (Part 1) or Day 1 to 92 for CNTO 3649 30 and 100 mcg/kg (Part 2)
  Area Under the Concentration-time Curve From Zero to Infinity (AUC [0 - infinity]) will be observed.
Apparent Systemic Clearance (CL/F) | Day 1 to 57 for CNTO 3649 10, 30, 100 and 300 mcg/kg (Part 1) or Day 1 to 92 for CNTO 3649 30 and 100 mcg/kg (Part 2)
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after subcutaneous dose (apparent systemic clearance) is influenced by the fraction of the dose absorbed (bioavailability).
Apparent Volume of Distribution (Vz/F) | Day 1 to 57 for CNTO 3649 10, 30, 100 and 300 mcg/kg (Part 1) or Day 1 to 92 for CNTO 3649 30 and 100 mcg/kg (Part 2)
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of a drug. Apparent volume of distribution after subcutaneous dose (Vz/F) is influenced by the fraction absorbed.
Mean Percentage Change From Baseline in Blood Glucose Values, Serum Insulin Concentration, and Serum C-Peptide Concentration | Day 1 to 57 for CNTO 3649 10, 30, 100 and 300 mcg/kg (Part 1) or Day 1 to 92 for CNTO 3649 30 and 100 mcg/kg (Part 2)
  Mean percentage change from baseline in blood glucose values, serum insulin concentration, and serum c-peptide concentration will be observed.
Weighted Average Blood Glucose (WAG) Level | Day -1 (Predose) and 24
  The WAG level is calculated as: WAG = Area under concentration (AUC) 24 /24 hours) the day before the first injection and on treatment Day 24 for CNTO 3649 30 or 100 mcg/kg for part 2 participants.
Change From Baseline in Glycosylated Haemoglobin (Hb) A1c at Day 36 and 50 | Baseline, Day 36 and 50
  Change From Baseline in Glycosylated Haemoglobin (Hb) A1c at Day 36 and 50 will be observed.
Number of Participants Exhibiting Anti-Drug Antibodies for CNTO 3649 at any Visit | Day 1 to 57 for CNTO 3649 10, 30, 100 and 300 mcg/kg (Part 1) or Day 1 to 92 for CNTO 3649 30 and 100 mcg/kg (Part 2)
  Number of participants exhibiting anti-drug antibodies for CNTO 3649 will be observed.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (1):
- Fukukoka, Japan

REFERENCES:
- See also: Safety, Pharmacokinetics, and Pharmacodynamics of a Single Subcutaneous Dose of CNTO 3649 in Healthy Adult Men and Multiple Subcutaneous Doses of CNTO 3649 in Patients With Type 2 Diabetes Mellitus — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=2352&filename=CR016429_CSR.pdf